CLINICAL TRIAL: NCT01269281
Title: Open Label, Randomized, Two Way Crossover, Comparative Evaluation of Relative Bioavailabilities of Two Formulations of Sumatriptan Succinate Tablets 100 mg (Dr. Reddy's Laboratories Limited, India)With the Reference Formulation Imitrex Tablets 100 mg (Glaxosmilthkine) in Healthy Adult Subjects Under Fed Conditions.
Brief Title: Bioequivalence Study of Sumatriptan Succinate Tablets 100 mg in Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: General Manager - Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BA0559019
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2005-10

CONDITIONS: Healthy
Keywords: Bioequivalence; two way crossover
MeSH Terms: interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sumatriptan Succinate tablets 100 mg (Experimental): Sumatriptan Succinate tablets 100 mg of Dr.Reddy's Laboratories Limited
  Interventions: Drug: Sumatriptan
- Imitrex 100 mg Tablets (Active Comparator): Imitrex 100 mg Tablets of Glaxosmithkline
  Interventions: Drug: Sumatriptan

INTERVENTIONS:
Drug: Sumatriptan — Sumatriptan Succinate Tablets 100 mg
  Other Names: Imitrex

SUMMARY:
The objective of this study was to compare the relative bioavailability of Sumatriptan Succinate Tablets 100 mg with Imitrex Tablets 100 mg under fed conditions in healthy adult human subjects.

DETAILED DESCRIPTION:
Open Label, Randomized, Two way crossover, comparative evaluation of relative bioavailability of two formulations of Sumatriptan Succinate Tablets 100 mg (Dr. Reddy's Laboratories Limited, India) With the Reference Formulation Imitrex® 100 mg Tablet (Glaxosmithkline, USA)Under Fed Conditions in Healthy Human Adult Subjects. 50 healthy, adult, human male subjects were enrolled in the study and 43 subjects are completed the study.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects should be healthy males between 18 and 45 years.
2. The subjects should be screened within 21 days prior to the administration of first dose of the study..
3. The subjects should have a BMI between 18 and 25 kg/m2
4. The subjects should be able to communicate effectively with study personnel
5. The subjects should be literate and able to give consent
6. If subject is a female volunteer and

   * Is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device(IUD), or abstinence
   * Is postmenopausal for at least 1 year
   * Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject).

Exclusion Criteria:

1. The subjects who have a history of allergic responses to Sumatriptan or other related drugs
2. The subjects who have history of intake of MAOI within two weeks of dosing
3. The subjects who have history of drug dependence, recent history of alcoholism or of moderate alcohol uses..
4. The subjects who have significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, ECG, and X-ray recordings..
5. The subjects who have any disease or condition which might compromise the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system, diabetes, psychosis or glaucoma or any other body system.
6. The subjects who have a history or presence of asthma (including aspirin induced asthma) or nasal polyp..
7. The subjects who are smokers and who smoke more than 10 cigarettes/day or those who cannot refrain from smoking during study period..
8. The subjects with a history of difficulty with donating blood or difficulty in accessibility of veins..
9. The subjects who have donated 01 unit (350 ml / 450 ml) blood within 90 days prior to receiving the first dose of study medication (if blood loss is below or equal to 200mL, subjects can be enrolled in the trial after 60 days of donation).
10. The subject who has a positive hepatitis screen including hepatitis B surface antigen, anti HCV, anti HEV.
11. The subject who has a positive test result for HIV antibody and / or syphilis (RPR/VDRL).
12. The subject who receives an investigational product, or has participated in a drug research study within a period of 90 days prior to the first dose of the study medication administration (elimination half-life of study drug should be taken into consideration for inclusion of subject in the trial if blood loss is below or equal to 200 mL).
13. An unusual diet, for whatever reason (e .g. low sodium) for four weeks prior to receiving the study medication and throughout the subject's participation in the study.
14. Female volunteers demonstrating a positive pregnancy screen.
15. Female volunteers who are currently breast- feeding.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2005-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUCt and AUCi parameters | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Roma Choudhury, MBBS, Principal Investigator — BA Research India Limited
Locations (1):
- BA Research India Limited, Bodakdev, Ahmedabad, India